CLINICAL TRIAL: NCT06256315
Title: Hyper Enhanced Recovery After Surgery (Hyper-ERAS) Program for Highly Selective Colorectal Cancer Patients Undergoing Laparoscopic Surgery
Brief Title: Hyper-ERAS Program for Highly Selective Colorectal Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Lin Wang, Unit III & Ostomy Service, Gastrointestinal Cancer Center, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PKUCH Hyper-ERAS research
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer; ERAS
Keywords: Colorectal Cancer; Hyper-ERAS; Super Accelerated Rehabilitation Surgery; Rapid Rehabilitation; Perioperative Management; ERAS2.0
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A:Hyper-ERAS(Length of Postoperative Hospital Stay<48h) (Experimental): Patients treated with the Hyper-ERAS rehabilitation protocol and discharged within 48 hours were in group A.
  Interventions: Procedure: Hyper-ERAS Program
- Group B:Hyper-ERAS(LOPS>48h) (Experimental): Patients treated with the ERAS rehabilitation protocol and discharged in more than 48 hours were in group B.
  Interventions: Procedure: Hyper-ERAS Program
- Group C:Control group (No Intervention): Patients eligible but not treated with the Hyper-ERAS rehabilitation protocol during the same period were in group C.

INTERVENTIONS:
Procedure: Hyper-ERAS Program — Patients who met the inclusion criteria were treated with Hype-ERAS protocol, including preoperative education, intraoperative quality control, postoperative preventive analgesia, early ambulation, early recovery of diet, early removal of the drainage tube, urinary catheter, and gastric tube, and discharge within 48 hours or more than 48 hours safter surgery, and closely and standardized follow-up outside the hospital.
  Arms: Group A:Hyper-ERAS(Length of Postoperative Hospital Stay<48h); Group B:Hyper-ERAS(LOPS>48h)

SUMMARY:
This clinical trial aims to explore the safety and effectiveness of the Hyper-ERAS rehabilitation protocol for colorectal cancer patients and the feasibility of discharge within 48 hours.

DETAILED DESCRIPTION:
The Hype-ERAS protocol includes preoperative education, intraoperative quality control, postoperative preventive analgesia, early ambulation, early recovery of diet, early removal of drainage tube, urinary catheter, and gastric tube, discharge within 48 hours after surgery, and standardized follow-up outside the hospital. Patients treated with the Hyper-ERAS rehabilitation protocol and discharged within 48 hours were in group A. Patients who were treated with Hyper-ERAS protocol and had a postoperative hospital stay of more than 48 hours were classified as group B. Patients eligible but not treated with the Hyper-ERAS rehabilitation protocol during the same period were in group C (Control group). The postoperative recovery of each group was compared to explore the safety and efficacy of Hyper-ERAS rehabilitation program in patients with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed colorectal cancer.
2. The position of the anastomosis is above the peritoneal reflection.
3. Age range from 18 to 79 years old.
4. No surgical contraindications.
5. The patient has good compliance and can understand the concept of rapid recovery.
6. Possess basic nursing conditions outside the hospital, and can arrive at the hospital within 30 minutes after discharge.

Exclusion Criteria:

* The exclusion criteria consisted of three parts: the first exclusion at enrollment, the second exclusion after surgery, and the third exclusion before discharge, corresponding to three exclusion criteria. 1st: Exclusion criteria at enrollment: 1). ASA grade ≥ grad 4. 2). Having previous surgical history, complex surgery, or combined/multiple organ resection with large trauma. 3). patients with complete obstruction or obvious intestinal edema and dilatation. 4). application of high-dose hormones, immunosuppressants, and preoperative radiotherapy. 5). Emergency surgery. 6). Patients with self-care difficulties for physical or mental reasons. 7). Pregnant patients. 8). to accept other studies simultaneously. 9). Inability to understand or accept the concept of enhanced recovery after surgery; 2nd: Postoperative exclusion criteria: 1). Adverse events occurred during preoperative preparation, such as perforation, massive bleeding, obstruction, fever, etc. 2). Adverse events occurred during the operation, such as intraoperative massive bleeding (≥400ml), unsatisfactory anastomosis, intraoperative perforation, unstable vital signs, etc. 3). Have any other conditions deemed ineligible for enrollment; 3rd: Exclusion criteria before discharge: 1). Body temperature above 37.5℃. 2) The food intake cannot meet the basic physiological needs, such as liquid food < 1000ml/ day. 3) with obvious abdominal distension, vomiting, cough and expectoration, dizziness, chest tightness, and other discomfort. 4) patients with abnormal laboratory indicators and abnormal nature of drainage fluid requiring hospitalization, such as bleeding, infection, leakage, etc. 5). Poor recovery of field activities and inability to care for themselves. 6). Have any other conditions deemed unsuitable for discharge. 7). Refusal to discharge.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
30-day overall complication rate | 30 days after surgery
  The primary endpoint was the 30-day overall complication rate.

SECONDARY OUTCOMES:
Severe complications (CD≥IIIb) rate, within 30 days after surgery | 30 days after surgery
  Severe complications (CD≥IIIb) rate
The rehospitalization rate within 30 days after surgery | 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Haidian District, China